CLINICAL TRIAL: NCT02120911
Title: Feasibility Study of Chemoradiation, TRAstuzumab and Pertuzumab in Resectable HER2+Esophageal Carcinoma: the TRAP Study
Brief Title: Feasibility Study of Chemoradiation, TRAstuzumab and Pertuzumab in Resectable HER2+ Esophageal Carcinoma
Acronym: TRAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, MD, PhD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCMEDONC 2013-377; 2013-004111-42 (EudraCT Number)
Record Dates: First submitted 2014-04-15; First posted 2014-04-23 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Esophageal Carcinoma
Keywords: Her2+; Resectable esophageal carcinoma; Pertuzumab; Trastuzumab
MeSH Terms: conditions — Esophageal Neoplasms | interventions — pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pertuzumab, trastuzumab (Experimental): Pertuzumab, trastuzumab
  Interventions: Drug: Pertuzumab, trastuzumab

INTERVENTIONS:
Drug: Pertuzumab, trastuzumab — Pertuzumab and trastuzumab will be combined with standard chemoradiation with carboplatin and paclitaxel.
  Other Names: Perjeta; Herceptin

SUMMARY:
Despite neoadjuvant chemoradiation regimens esophageal cancer remains a disease with poor outcome. The clinical benefit of HER2 targeting with trastuzumab has been shown in the setting of advanced disease and disease and safety of combining trastuzumab with chemoradiation in the curative setting has been established. In breast cancer, the added value of pertuzumab to standard treatment with trastuzumab has been shown both in the neoadjuvant and the metastastic setting. Taken together, there is a sound rationale to explore the combination of radiotherapy plus chemotherapy with trastuzumab and pertuzumab in HER2+resectable esophageal cancer. However, since the number of HER2+ patients in this setting is limited, and no data are available on the safety of this combination prior to major surgery, we propose to first conduct a feasibility study with this treatment stratgy. When the results of this study show that this treatment strategy is feasible, we will subsequently design a prospective study with efficacy as primary endpoint.

DETAILED DESCRIPTION:
Objective of the study:

Assess the feasibility of preoperative treatment with pertuzumab and trastuzumab combined with preoperative chemoradiation (carboplatin, paclitaxel and radiation) in terms of withdrawal rate from surgery.

Study design:

This is a non-randomized feasibility study with Paclitaxel (T), Carboplatin (C), Pertuzumab (P). Trastuzumab (H), and radiation (RT) followed by surgical resection of the oesophagus.

Study population:

Patients (male/female) with histologically proven adenocarcinoma of the intrathoracic esophagus or gastro esophageal junction, age >18 and <75 years.

Intervention (if applicable):

Paclitaxel 50 mg/m2 and Carboplatin AUC = 2 will be given by intravenous infusion on days 1, 8, 15, 22 and 29.

Trastuzumab will be administered at a dose of 4 mg/kg on day 1, followed by 2 mg/kg at wk 2-6. From wk 7 onwards trastuzumab is administered at a dose of 6 mg/kg every 3 weeks. Pertuzumab will be given 840 mg intravenously at each administration.

Thus, trastuzumab and pertuzumab will be continued during eight weeks after the end of chemoradiation. Surgery will be planned in or around week 14, approximately eight weeks after the end of chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the intrathoracic esophagus or gastro esophageal junction.
* HER2-positive tumor defined as either IHC 3+ or IHC 2+, the latter in combination with ISH+, as assessed by the sponsor-designated central laboratory (pathology AMC) on a primary tumor biopsy.
* Surgical resectable (T2-3, N0-1, M0), as determined by Endoscopic Ultra Sound (EUS) and CT scan of neck, thorax and abdomen.
* T1N1 tumors are eligible, T1N0 tumors and in situ carcinoma are not eligible.
* Tumor length longitudinal ≤ 10 cm and radial ≤ 5 cm.
* If tumor extends below the gastroesophageal (GE) junction into the proximal stomach, the bulk of the tumor must involve the esophagus or GE junction. The tumor must not extend more than 2 cm into the stomach.
* No invasion of the tracheobronchial tree or presence of tracheoesophageal fistula.
* Age ≥ 18 and ≤ 75 years.
* ECOG performance status 0 or 1.
* Adequate hematological, renal and hepatic functions defined as:

  * neutrophiles ≥ 1.5 x 109/L
  * platelets ≥ 100 x 109/L
  * hemoglobin ≥ 5.6 mmol
  * total bilirubin ≤ 1.5 x upper normal limit
  * creatinine clearance (Cockroft) > 60 ml/min
* Adequate left ventricular ejection fraction defined as an LVEF of ≥55%.
* Written, voluntary informed consent.
* Patients must be accessible to follow up and management in the treatment center.

Exclusion Criteria:

* A tumour the epicenter of which in the stomach is greater than 5 cm of the GE junction or those within 5 cm of the GE junction without extension in the oesophagus are classified as gastric cancer.
* Past or current history of malignancy other than entry diagnosis except for non-melanomatous skin cancer, or curatively treated in situ carcinoma of the cervix, or malignancy more than 5 years prior to enrollment.
* Pregnancy (positive serum pregnancy test), planning to become pregnant, and lactation.
* Patient (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.
* Previous chemotherapy, radiotherapy, treatment with an anti-HER2 antibody or with small molecule HER2 inhibitors.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before randomization.
* Pulmonary fibrosis and/or severely impaired lung function.
* Pre-existing motor or sensory neurotoxicity greater than WHO grade 1.
* Active infection or other serious underlying medical condition which would impair the ability of the patient to receive the planned treatment, including prior allergic reactions to drugs containing Cremophor, such as teniposide or cyclosporine.
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent
* Inadequate caloric- and/or fluid intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
% of patients completing trastuzumab and pertuzumab treatment. | up to 14 weeks after start of treatment
  See title

SECONDARY OUTCOMES:
Toxicity of pertuzumab and trastuzumab alone and in combination with chemoradiation | up to 14 weeks after start of treatment
  See title
Number of post-operative complications | up to 3 months after surgery
  See title
Pathological response | up to 2 weeks after surgery
  See title
R0 resection rate | up to 2 weeks after surgery
  See title
Pharmacokinetics of pertuzumab and trastuzumab | up to 14 weeks after start of treatment
  See title

OTHER OUTCOMES:
Relation between exposure and effect (safety and efficacy). | up to 3 months after surgery
  See title
Biomarker analyses | up to 3 months after surgery
  See title
SUV of pre-treatment trastuzumab-PET | up to two weeks after surgery
  See title

CONTACTS AND LOCATIONS:
Overall Officials: H. WM van Laarhoven, MD, PhD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Medical Oncology, Amsterdam, Netherlands

REFERENCES:
- [Result] Stroes CI, Schokker S, Creemers A, Molenaar RJ, Hulshof MCCM, van der Woude SO, Bennink RJ, Mathot RAA, Krishnadath KK, Punt CJA, Verhoeven RHA, van Oijen MGH, Creemers GJ, Nieuwenhuijzen GAP, van der Sangen MJC, Beerepoot LV, Heisterkamp J, Los M, Slingerland M, Cats A, Hospers GAP, Bijlsma MF, van Berge Henegouwen MI, Meijer SL, van Laarhoven HWM. Phase II Feasibility and Biomarker Study of Neoadjuvant Trastuzumab and Pertuzumab With Chemoradiotherapy for Resectable Human Epidermal Growth Factor Receptor 2-Positive Esophageal Adenocarcinoma: TRAP Study. J Clin Oncol. 2020 Feb 10;38(5):462-471. doi: 10.1200/JCO.19.01814. Epub 2019 Dec 6. PMID 31809243